CLINICAL TRIAL: NCT03966963
Title: A Systematic Case Series Study Investigating the Effectiveness of Eye Movement Desensitization Reprocessing (EMDR) in the Treatment of Childhood Sexual Abuse in Adolescents and Adult Survivors
Brief Title: Systematic Case Series Investigating Eye Movement Desensitization Reprocessing (EMDR) Efficacy With Childhood Sexual Abuse Survivors
Acronym: EMDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salford (Other)
Responsible Party: Principal Investigator, Halima Bibi, Postgraduate Research Student, University of Salford
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 786
Record Dates: First submitted 2019-05-22; First posted 2019-05-29 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Trauma, Psychological
Keywords: Eye Movement Desensitization Reprocessing; EMDR; childhood sexual abuse; posttraumatic stress disorder; PTSD; adults
MeSH Terms: conditions — Psychological Trauma; Stress Disorders, Post-Traumatic | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Intervention Model Description: Mixed methods study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eye Movement Desensitization Reprocessing (EMDR) (Experimental): Subjects with trauma-related symptomology resultant from CSA will undertake EMDR; they will be systematically observed through use of their quantitative treatment outcome measures at both pre- and post- treatment alongside one-month follow-up interview data to determine outcomes of interest (namely emotional, behavioural and neuropsychological functioning).
  Interventions: Behavioral: Eye Movement Desensitization Reprocessing (EMDR)

INTERVENTIONS:
Behavioral: Eye Movement Desensitization Reprocessing (EMDR) — Trauma-Focused Therapy

SUMMARY:
This study investigates the effectiveness of EMDR for survivors of childhood sexual abuse. All participants will undertake a standard course of EMDR via the National Heath Service program, alongside a number of questionnaires and a follow-up interview.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effectiveness of Eye Movement Desensitisation Reprocessing (EMDR) via investigation of the changes in the individual trauma stress response on sexually abused adolescents and young adults, aged between 18 and 25 during EMDR treatment. The findings of this mixed methods study will explore (a) neuropsychological, emotional (namely low self-esteem, anxiety and depression), behavioural functioning and quality of life issues via quantitative measures conducted before, during and after treatment and (b) client perspectives of such changes through qualitative interviewing (interview guide is in Appendix 7) at one month follow-up using Interpretative Phenomenological Analysis [IPA]. The study setting will be conducted within the Improving Access to Psychological Therapies (IAPT) program framework, established to ensure service users accessing NHS treatment are presented with choice in their treatment. Therapy will routinely be delivered within GP Surgeries or Health Centres.

Within this two-fold study, the following key research questions will be considered in relation to the effectiveness of EMDR:

1. Qualitative data will sought to identify; In what ways was EMDR helpful? In what ways was EMDR perceived as being unhelpful?
2. Quantitative data will sought to identify; Are there changes in emotional and behavioural functioning (in relation to trauma, anxiety and depressive symptoms)? Are there changes in neuropsychological functioning (memory, attention, executive functioning)? Are there changes in quality of life issues? Are there changes in self-worth?

ELIGIBILITY:
Inclusion Criteria:

Participants, both male and female, aged between 18 and 25, whom;

* have experienced CSA before the age of 16
* exhibit PTSD symptomology
* ensure PTSD symptomology is present for over three-months and primarily derived from pre-16 aged trauma
* be available for treatment-sessions on a weekly basis for up to 16-sessions - have good understanding of the English language to avoid language barriers/additional time spent with interpreters
* if taking medication, this will have been stable for a period of at least 2-months prior to therapy
* EMDR is the sole treatment for PTSD from baseline until follow-up to avoid conflict of interest

Exclusion Criteria:

Participants exhibiting;

* significant psychiatric comorbidity
* comorbid psychotic disorder
* bipolar disorder type 1
* alcohol or drug dependence
* acute suicide risk, acute PTSD from trauma within the past 6 months
* PTSD focused treatment within the past 3 months or scheduled to begin another form of PTSD treatment will be excluded
* those currently participating in research or have recently participated in conflicting research

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Impact of Events Scale-Revised 'IESR' | Change from Baseline PTSD symptomology at up to 5 months
  22-item self-report measure to evaluate impact of sexual abuse in terms of traumatic stress, abuse attributions and social reactions. Participants will be asked to rate their level of distress in relation to the said traumatic event on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"), ultimately providing the researcher with a total score (ranging from 0 to 88). The higher the score, the greater the PTSD symptomology.
The Psychology Experiment Building Language 'PEBL' Test | Change from Baseline neuropsychological functioning at up to 5 months
  The PEBL is an electronic neuropsychological battery utilised to monitor adaptations in participants' neuropsychological functioning.
Generalized Anxiety Disorder 7 (GAD-7) Scale | Change from Baseline anxiety levels at up to 5 months
  Participants will be asked to rate their level of anxiety on a 7-point scale ranging from 0 ("not at all") to 3 ("nearly every day"), ultimately providing the researcher with a total score (ranging from 0 to 21). The higher the score, the greater the anxiety.
Patient Health Questionnaire 9 (PHQ-9) Scale | Change from Baseline depression levels at up to 5 months
  Participants will be asked to rate their level of depression on a 9-point scale ranging from 0 ("not at all") to 3 ("nearly every day"), ultimately providing the researcher with a total score (ranging from 0 to 27). The higher the score, the greater the depression.
Weekly Problems Rating Scale | Change from Baseline emotional and behavioural functioning at up to 5 months
  This consists of 11 statements that participants are requested to rate in order to describe their feelings and interactions during the past week to gauge general emotional and behavioural functioning. Answers/statements for all questions are from a choice of the following "never" "almost never" "a little of the time" "some of the time" "most of the time" "all of the time." Generally, the more negative the selected statement, the greater the indication of issues in functioning within that given domain.
Rosenberg Self-Esteem Scale 'RSES' | Change from Baseline levels of self-worth at up to 5 months
  The 10-item RSES measures global self-worth by measuring both positive and negative feelings about the self. Participants will be asked to rate their level of self-worth by measuring both positive and negative feelings about the self. All items are answered using a 4-point Likert scale format as follows; "Strongly Disagree" 1 point, "Disagree" 2 points, "Agree" 3 points, and "Strongly Agree" 4 points,' ultimately providing the researcher with a total score (ranging from 10 to 40). Higher scores indicate higher self-esteem.
The Valued Living Questionnaire 'VLQ' | Change from Baseline quality of life issues at up to 5 months
  The VLQ is an instrument that taps into 10 valued domains of living as follows; 1. Family, 2. Marriage/couples/intimate relations, 3. Parenting, 4. Friendship, 5. Work, 6. Education, 7. Recreation, 8. Spirituality, 9. Citizenship, and 10. Physical self-care. Scoring: Respondents are asked to rate the 10 areas of life on a scale of 1 (not at all important) -10 (extremely important), indicating the level of importance and how consistently they have lived in accord with those values in the past week, ultimately providing the researcher with a total score (ranging from 10 to 100).

SECONDARY OUTCOMES:
Helpful Aspects of Therapy Interview | One-month follow up
  A qualitative semi-structured interview at one-month follow up. The first seven questions of which will help identify helpful/unhelpful aspects of therapy and the final four questions focusing on effectiveness, ending and any recommendations for treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Dubrow-Marshall, Study Chair — University of Salford; Clare S Allely, Study Chair — University of Salford
Locations (1):
- Greater Manchester Mental Health NHS Trust (GMMH - IAPT Headquarters, Chorlton House), Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This study forms part of a doctorate qualification, as per University policy, all data will comply will GDPR (2018) and may be stored on a University encrypted drive for up to three years. The thesis itself may contain non-identifiable patient data such as interview extracts however this will be limited to consent.

REFERENCES:
- [Derived] Brown SJ, Carter GJ, Halliwell G, Brown K, Caswell R, Howarth E, Feder G, O'Doherty L. Survivor, family and professional experiences of psychosocial interventions for sexual abuse and violence: a qualitative evidence synthesis. Cochrane Database Syst Rev. 2022 Oct 4;10(10):CD013648. doi: 10.1002/14651858.CD013648.pub2. PMID 36194890